CLINICAL TRIAL: NCT07032506
Title: A Randomized Controlled Trial of Intrauterine Stent Placement Following Hysteroscopic Septum Resection
Brief Title: Intrauterine Stent Placement Following Hysteroscopic Septum Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-04027291
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Intrauterine Adhesion
Keywords: intrauterine foley balloon catheter stent; uterine malformations; uterine septums; hysteroscopic septoplasty
MeSH Terms: conditions — Gynatresia; Uterine Anomalies; Septate Uterus | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention A:Intraoperative placement of an inflated intrauterine pediatric foley catheter (Experimental): Intraoperative placement of an inflated intrauterine pediatric foley catheter balloon to remain in place for 7-10 days following surgery.
  Interventions: Procedure: Intraoperative placement of an inflated intrauterine pediatric foley catheter; Drug: Hormonal Therapy Agent; Drug: Oral antibiotics
- Intervention B: No placement of placement of an inflated intrauterine pediatric foley catheter (Active Comparator): No placement of an inflated intrauterine pediatric foley catheter
  Interventions: Procedure: No Catheter placement; Drug: Hormonal Therapy Agent

INTERVENTIONS:
Procedure: Intraoperative placement of an inflated intrauterine pediatric foley catheter — Intraoperative placement of an inflated intrauterine pediatric foley catheter balloon to remain in place for 7-10 days following surgery.
  Arms: Intervention A:Intraoperative placement of an inflated intrauterine pediatric foley catheter
Procedure: No Catheter placement — No Intraoperative placement of an inflated intrauterine pediatric foley catheter balloon
  Arms: Intervention B: No placement of placement of an inflated intrauterine pediatric foley catheter
Drug: Hormonal Therapy Agent — 2 weeks of oral estradiol (2 mg daily) or transdermal (two 0.1 mg patches changed twice weekly) estradiol supplementation followed by 1 week of oral or transdermal estradiol (same dosing as above) with oral medroxyprogesterone acetate (10 mg daily)
Drug: Oral antibiotics — 100 mg of oral doxycycline twice daily or other appropriate antibiotic in allergic patients to be given while the intrauterine stent is in place
  Arms: Intervention A:Intraoperative placement of an inflated intrauterine pediatric foley catheter

SUMMARY:
The study hopes to learn the best way to prevent internal scar tissue after septum removal. The use of an intrauterine foley catheter balloon may prevent the formation of adhesions following surgery.

DETAILED DESCRIPTION:
This is an open label randomized controlled clinical trial of post-operative interventions to prevent intrauterine adhesion formation following hysteroscopic septoplasty. Individuals undergoing planned hysteroscopic resection of a known uterine septum with a length of ≥50% of the uterine cavity, as measured from the lower uterine segment to the inter-cornual line on 3D ultrasound or MRI will be randomized to either placement of an intrauterine foley catheter balloon for 7-10 days with hormonal supplementation or hormonal supplementation only. Individuals unwilling or unable to consent, those with a history of prior transmural uterine surgery, those with a history of a prior septum resection, history of prior surgery for intrauterine adhesions, or individuals in whom complete septum resection is unable to be performed in a single procedure will be excluded.

Patients will be screened by study investigators for eligibility. Patients will be identified if they are found to have a uterine septum during their evaluation for infertility or recurrent pregnancy loss or if previously identified by a referring provider. Investigators will obtain written informed consent in the patient's preferred language by person-to-person contact. Patients choosing to enroll will be randomized in a 1:1 allocation to one of two interventions:

Surgical technique in the form of electrocautery versus sharp resection will be at the surgeon's discretion. All patients will undergo a post-operative in-clinic 3D saline sonogram to assess adhesion formation within the first two menstrual cycles following the intervention, to be performed no later than 12 weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Patients electing to undergo hysteroscopic septoplasty following an informed consent and shared decision making process
* Uterine septum of at least 50% of the uterine cavity length as quantified on 3-dimensional saline infusion ultrasound

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* History of prior uterine septum resection
* History of prior transmural uterine surgery
* Preexisting intrauterine adhesions or prior treatment for intrauterine adhesions
* Individuals in whom complete septum resection is unable to be performed as a single procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of intrauterine adhesion formation following hysteroscopic septoplasty | 12 weeks

SECONDARY OUTCOMES:
Number of participants with Intraoperative complications | 12 weeks
Number of participants with postoperative complications | 12 weeks
Number of subjects completing postop intervention-hormone use | 12 weeks
Patient compliance - Post Operative - #subject with balloon remaining in place to post op visit | 12 weeks
Long Term Reproductive Outcome | 3 years
  Number of subjects achieving pregnancy
Surgeon assessment of intervention modality | 12 weeks
  Surgeon assessment of whether intrauterine adhesions were prevented

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Schattman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Arkansas Fertility & Gynecology, Little Rock, Arkansas
  - Weill Cornell Medicine, New York, New York
  - University Hospitals, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No